CLINICAL TRIAL: NCT04729478
Title: Comparison Between Natural Sleep Endoscopy and Drug-induced Sleep Endoscopy in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ethisch.comite@uza.be (Other)
Responsible Party: Sponsor-Investigator, ethisch.comite@uza.be, Olivier Vanderveken, Professor and Chair Otorhinolaryngology, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: B3002021000006
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea; Sleep Apnea Syndromes; Apnea; Respiration Disorder; Respiratory Tract Disease; Dyssomnia; Sleep Disorders, Intrinsic; Sleep Wake Disorders; Nervous System Diseases; Hypnotics and Sedatives; Central Nervous System Depressants; Propofol; Midazolam; Physiological Effects of Drugs; General Anesthetics
Keywords: Sleep endoscopy; Sedation; Airflow analysis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Apnea; Respiration Disorders; Respiratory Tract Diseases; Dyssomnias; Sleep Disorders, Intrinsic; Sleep Wake Disorders; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Blinded, prospective, single-center, comparative cohort study.
Who Masked: Outcomes Assessor
Masking Description: NSE and DISE will be performed by two separate researchers, blinding the ENT surgeon who performs the NSE or DISE for the outcome of the other procedure. This is a blinded study and the researchers will have no knowledge of the patient's characteristics / demographic variables and their history.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural sleep (Other): Natural sleep endoscopy (NSE)
  OSA patients will be endoscopically evaluated during natural sleep.
  During NSE additional physiological measurements (flow shape analysis, acoustic analysis of snoring sounds and esophageal pressure measurements) will be carried out.
  Interventions: Device: Natural sleep endoscopy
- Drug-induced sleep (Other): Drug-induced sleep endoscopy (DISE)
  OSA patients will be endoscopically evaluated during drug-induced sleep.
  During DISE additional physiological measurements (flow shape analysis, acoustic analysis of snoring sounds and esophageal pressure measurements) will be carried out.
  Interventions: Device: Drug-induced sleep endoscopy

INTERVENTIONS:
Device: Drug-induced sleep endoscopy — An intravenous bolus injection of midazolam 1.5 mg will be used to induce sleep. Maintenance of sedated sleep will be obtained by a target-controlled infusion of propofol (2.0-3.0 µg/mL).
  Other Names: DISE
  Arms: Drug-induced sleep
Device: Natural sleep endoscopy — Endoscopy during natural sleep.
  Other Names: NSE
  Arms: Natural sleep

SUMMARY:
Drug-induced sleep endoscopy (DISE) is the most used technique for identifying the obstruction site associated with obstructive sleep apnea (OSA). This is due to the fact that it allows many patients to be examined in a daytime setting. This procedure uses sedative drugs to mimic natural sleep. However, associations with the site of upper airway (UA) collapse during natural sleep remain unclear.

The aim of this explorative study is to identify UA collapse in patients with OSA using endoscopic techniques as well as flow shape characteristics and sound analyses during natural and drug-induced sleep. Furthermore, we want to optimize the measurement set-up of natural sleep endoscopy (NSE).

DETAILED DESCRIPTION:
Patients with moderate to severe OSA requiring DISE will be recruited for this prospective study at the outpatient clinic. Patients will undergo a NSE at the sleep lab at night, and a DISE at the operating theatre within three months. Both the NSE and DISE set-up will include gold-standard flow measurements, acoustic analysis and esophageal pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA with a baseline AHI ≥ 15 per hour based on full polysomnography
* Body mass index (BMI) ≤ 35 kg/m²
* Capability of giving informed consent and willingness to undergo NSE

Exclusion Criteria:

* Central sleep apnea (defined as CAHI ≥ 30% of total AHI)
* Inability to sleep in a supine position due to a medical condition
* Inability of the patient to understand and/or comply to the study procedures
* Neuromuscular disorders or craniofacial anomalies affecting the UA
* Sedative medication use (opioids and muscle relaxants)
* Active psychiatric disorders (psychotic illness, major depression, anxiety attacks, excessive alcohol or drug use)
* Severe or decompensated cardiac or respiratory diseases
* Medical history of known causes of tiredness by day or severe sleep disruption (insomnia, PLMS, narcolepsy)
* Contra-indications for DISE: i.e. fitness for general anesthesia (ASA>3), allergy to sedative agent(s) and an expected extremely difficult airway
* Pregnancy or willing to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Endoscopic Classification System | Immediately, during the procedure
  Comparison of the frequencies of the site, gradation and pattern of upper airway collapse between natural and drug-induced sleep endoscopy.

SECONDARY OUTCOMES:
Flow shape analysis | Immediately, during the procedure
  Several parameters extracted from the flow signal, including negative effort dependence (NED), peak inspiratory flow, etc. measured during both natural and drug-induced sleep endoscopy.
Acoustic analysis | Immediately, during the procedure
  Acoustic analyses measured during both natural and drug-induced sleep endoscopy

OTHER OUTCOMES:
Apnea-hypopnea index (AHI) | Immediately, during polysomnography
  The AHI is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow).
Oxygen desaturation index (ODI) | Immediately, during polysomnography
  The ODI represents the average number of desaturation episodes (≥3%) per hour sleep.
Oxygen saturation (SaO2) | Immediately, during polysomnography
  Minimal and mean SaO2 (%)
Apnea index | Immediately, during polysomnography
  The apnea index is an index of sleep apnea severity that encompasses the frequency of apneas.
Arousal index | Immediately, during polysomnography
  The arousal index is an indirect indicator of sleep apnea severity that encompasses the number of arousals related to total sleep time.
Arousal threshold | Immediately, during polysomnography
  The occurrence of arousal from sleep with a rise in ventilatory drive.
Daytime sleepiness measured with the Epworth Sleepiness Scale (ESS) | Immediately, before the procedure
  The probability of falling asleep in various settings and situations in daily life will be assessed. This questionnaire consists of eight questions which can be scored on a four-point Likert-type scale. The lowest score (zero) suggests that the described incident is absent and the highest score (three) suggests the presence of this event. The summation of the eight items can range from 0 to 24.
Checklist Individual Strength questionnaire (CIS20R) for fatigue | Immediately, before the procedure
  The checklist individual strength (CIS20R) is a 20-item questionnaire to assess the degree of fatigue. The patient selects the most appropriate score on each statement ranging from 1 (yes, this is true) to 7 (no, this is not true). The total score, calculated as the sum of the questions, may yield to a maximum of 140. The CIS20R measures four dimensions of fatigue: fatigue severity (8 items), concentration problems (5 items), reduced motivation (4 items) and activity (3 items).
Snoring intensity measured with a Visual Analogue Scale (VAS) | Immediately, before the procedure
  The subjective degree of snoring during sleep will be evaluated by the partner of a subject by using a VAS scoring system ranging from 0 (no snoring) to 10 (extreme snoring causing the bed partner to sleep separately). Heavy snoring is determined as a snoring index ≥7.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Van den Bossche K, Van de Perck E, Wellman A, Kazemeini E, Willemen M, Verbraecken J, Vanderveken OM, Vena D, Op de Beeck S. Comparison of Drug-Induced Sleep Endoscopy and Natural Sleep Endoscopy in the Assessment of Upper Airway Pathophysiology During Sleep: Protocol and Study Design. Front Neurol. 2021 Dec 7;12:768973. doi: 10.3389/fneur.2021.768973. eCollection 2021. PMID 34950101